CLINICAL TRIAL: NCT03386890
Title: Clinical Application of Non-invasive Assessment for Staging Liver Steatosis and Liver Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jidong Jia, Chief Physician, Beijing Friendship Hospital
Other Study IDs: XMLX201606
Record Dates: First submitted 2017-12-06; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Nonalcoholic Fatty Liver Disease; Liver Steatosis; Liver Fibrosis
Keywords: Non-invasive Assessment; Transient Elastography; Controlled Attenuation Parameter
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — liver histological section
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nowadays, the morbidity of Nonalcoholic fatty liver disease (NAFLD) show ascending trend year by year, which has become an important public health problem in China. As NAFLD can progress to Non-alcoholic steatohepatitis (NASH), cirrhosis and Hepatocarcinoma, the identification and quantitative evaluation of liver steatosis and its dynamic changes are crucial. While liver biopsy is still the gold standard in the diagnosis of NAFLD, its application is limited because of the invasive procedure.The Transient Elastography(TE) combined with the Controlled Attenuation Parameter(CAP) is a new non-invasive diagnostic method for fatty liver and liver fibrosis.

In order to evaluate the diagnostic value of non-invasive assessment for the degree of liver steatosis and staging liver fibrosis, this non-invasive method will be assessed by the golden standard of liver biopsy among 400 NAFLD patients.The treatment protocols will be decided by doctor and patient both (treatment protocols and medicine are not required). Blood routine, blood biochemistry, abdominal ultrasound and Transient Elastography(TE) combined with the Controlled Attenuation Parameter(CAP) are detected during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age:18≤,≥65
* Gender:male or female
* NAFLD patient,agree with the paracentesis of liver tissue
* Regular follow-up
* Signing the Informed Consent Form

Exclusion Criteria:

* Hepatic decompensation：Including cirrhotic complications,such as ascites,hepatic encephalopathy,digestive tract bleeding,hepatorenal syndrome,spontaneous bacterial peritonitis,and HCC.
* Complications of HBV,HCV,HIV.Complications of alcoholic liver disease,autoimmune liver disease,hereditary metabolic liver disease, drug-induced liver disease and other chronic liver disease.
* AFP>100ng/ml and imaging indicates malignant occupying.Or AFP still>100ng/ml within 3 months.
* Creatinine was 1.5 times higher than the upper limit of the normal value.
* Combined with other malignant tumors(except those cured).
* Serious diseases of heart, lung, kidney, brain, blood and other important organs with dysfunction.
* severe neurological and psychiatric diseases (such as epilepsy, depression, mania, schizophrenia, etc.)
* Pregnant women and breast-feeding women.
* The researchers consider that it is not suitable for the patients to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NAFLD male or female patints from 18 to 65 years old,who agree with the paracentesis of liver tissue and agree to sign the informed consent form.They are accessible for regular follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver Biopsy | 1 year
  liver histological section
CAP | 1 year
  Controlled Attenuation Parameter
TE | 1 year
  Transient Elastography

SECONDARY OUTCOMES:
Blood routine test | 1 year
  Blood routine test
liver biochemistry test | 1 year
  liver biochemistry test
abdominal ultrasound | 1 year
  abdominal ultrasound
electrolyte | 1 year
  electrolyte
blood glucose | 1 year
  blood glucose
blood lipid | 1 year
  blood lipid
uric acid | 1 year
  uric acid
kidney function test | 1 year
  kidney function test

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tong X, Sun Y, Wang Q, Zhao X, Chen W, Zhang M, Ren Y, Zhao X, Wu X, Zhao J, Sun C, Zheng M, Ren H, Yang Z, Ou X, Jia J, You H. Delicate and thin fibrous septa indicate a regression tendency in metabolic dysfunction-associated steatohepatitis patients with advanced fibrosis. Hepatol Int. 2025 Feb;19(1):166-180. doi: 10.1007/s12072-024-10719-w. Epub 2024 Aug 16. PMID 39152361
- [Derived] Wang Q, You H, Ou X, Zhao X, Sun Y, Wang M, Wang P, Wang Y, Duan W, Wang X, Wu S, Kong Y, Saxena R, Gouw ASH, Jia J. Non-obese histologically confirmed NASH patients with abnormal liver biochemistry have more advanced fibrosis. Hepatol Int. 2019 Nov;13(6):766-776. doi: 10.1007/s12072-019-09982-z. Epub 2019 Sep 26. PMID 31559605